CLINICAL TRIAL: NCT01729026
Title: A Study of Dog Adoption in Veterans With Posttraumatic Stress Disorder
Brief Title: A Study of Dog Adoption in Veterans With Posttraumatic Stress Disorder (PTSD)
Acronym: VITAL
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D0809-P
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: Veterans; Posttraumatic Stress Disorder; dog adoption; companion animal
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shelter Dog Adoption (Experimental): Veterans will choose a dog from the San Antonio Humane Society with the help of a Humane Society adoption counselor and study staff and take it home to live with them. The dog will be a pet and not a service dog. Following adoption, Veterans and their dogs will receive eight weeks of free obedience training provided by a veterinarian.
  Interventions: Other: Shelter Dog Adoption
- Wait-list, Then Adoption after 3 Months (Active Comparator): After 3 months on a wait-list, Veterans will choose a dog from the San Antonio Humane Society with the help of a Humane Society adoption counselor and study staff and take it home to live with them. The dog will be a pet and not a service dog. Following adoption, Veterans and their dogs will receive eight weeks of free obedience training provided by a veterinarian.
  Interventions: Other: Shelter Dog Adoption

INTERVENTIONS:
Other: Shelter Dog Adoption — Veterans will choose a dog from the San Antonio Humane Society with the help a Humane Society adoption counselor and study staff and take it home to live with them. The dog will be a pet and not a service dog. Following adoption, Veterans and their dogs will receive eight weeks of free obedience training provided by a veterinarian.

SUMMARY:
The purpose of this study is to provide preliminary data on the feasibility and impact of adopting a dog from an animal shelter as a supplement to usual care in Veterans with Posttraumatic Stress Disorder (PTSD) who desire to get such a pet.

DETAILED DESCRIPTION:
Posttraumatic Stress Disorder, a common mental disorder among Veterans, is marked by painful re-experiencing of a traumatic event, often together with depression, fearfulness, and social isolation. Despite major advances in rehabilitation, many Veterans continue to be disabled by PTSD. One possible new approach involves the use of shelter dogs, which might relieve symptoms and aid reintegration into society by providing emotional support and a greater sense of security. In this randomized controlled trial of 48 Veterans with chronic PTSD, we will evaluate whether the half who adopt a dog from the San Antonio Humane Society show greater improvement in their PTSD symptoms over the first three months than the half who are assigned to a waiting list.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual for Mental Disorders, Fifth Edition (DSM-5) criteria for current PTSD as determined by the Clinician-Administered PTSD Scale for DSM-5 (CAPS)
* Scores 39 or greater on the PTSD Checklist for DSM-5 (PCL-5)
* Feels able to afford to care for a dog after the anticipated annual costs of approximately $750 are outlined
* If married or cohabiting, spouse or significant other agrees with the decision to adopt a dog
* If not a homeowner, landlady or landlord agrees to allow the dog to reside on the property
* Agrees to keep the dog inside most of the time
* Agrees to be the primary caretaker for the dog
* Had a dog previously as a child or adult
* Served during the Vietnam era or more recently
* In active therapy for at least 1 month, with plans to remain in active therapy
* Has been in a stable housing situation for the last 3 months
* Case manager for any Veteran who is in the Housing and Urban Development/VA Subsidized Housing (HUD/VASH) program has been consulted prior to study enrollment
* Has a plan for someone else to take care of the dog if she or he can't

Exclusion Criteria:

* Has had a dog or other companion animal within the past 12 months
* Has current alcohol or drug abuse or dependence
* Has a primary psychiatric diagnosis other than PTSD
* Has had significant suicide/homicide risk in the past 3 months
* Has had psychosis or mania in the past 3 months
* Has had a psychiatric admission during the past 3 months
* Has mental or physical impairments that would interfere with caring for the dog or self
* Has a history of moderate to severe traumatic brain injury (TBI) (subjects with moderate TBI will be allowed to participate in the study if a Physical Medicine and Rehabilitation physician determines it is acceptable)
* Requires a puppy
* Requires a breed that is uncommonly available for adoption at the San Antonio Humane Society
* Requires a pit bull or other fierce dog
* Veteran's mental health clinician or Physical Medicine and Rehabilitation physician reports a past history of animal cruelty or abuse or expresses concern about the potential for such behavior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L. Stern, MD BA, Principal Investigator — South Texas Health Care System, San Antonio, TX
Locations (1):
- South Texas Health Care System, San Antonio, TX, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment opened in October 2013 and closed at the end of September 2014. Subjects learned about the study primarily from clinical staff or from posters and brochures that were distributed throughout the clinics of the South Texas Veterans Health Care System in San Antonio.
Pre-assignment Details: Two of the 22 consented subjects were not randomized: one left before he was evaluated and the second did not meet entry criteria. A third subject was randomized to the Adoption group but subsequently found not to meet criteria for PTSD, leaving 9 in this group and 10 in the Wait-List group.
Period: Randomization to 3-month Follow-up
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months
Started | 9 | 10
Completed | 7 | 8
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2
Period: 3-month to 6-month (Final) Follow-up
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months
Started | 7 | 8
Completed | 6 | 6
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (13.8) | 39.2 (11.4) | 42.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Checklist (PCL-5) Score Between Baseline and 3-month Follow-up
Description: The PCL-5 is a self-rating scale based on the DSM-5 diagnostic criteria for Posttraumatic Stress Disorder. The range of the scale is from 0 (no symptoms) to 80 (maximal symptoms).
Time Frame: Baseline and 3-month follow-up visit.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months
Number analyzed (Participants) | 9 | 10
units on a scale | -15.20 (3.52) | -7.77 (3.29)
Statistical Analysis 1: Comparison: Shelter Dog Adoption vs Wait-list, Then Adoption After 3 Months; The analyses were mixed effect regression models with repeated measures at randomization (baseline) and at the 3-month post-randomization follow-up using a 2 x 2 design. Treatment (Adoption group vs Wait-list group), time (baseline and 3-month follow-up) and their interaction were the fixed design effects. The treatment by time interaction tests the significance of the difference between baseline and 3-month follow-up between the Adoption and Wait-list groups; Test type: Superiority or Other; p = 0.141, Mixed effects regression models — Between baseline and 3-month follow-up, subjects in the Adoption group had a mean improvement of 15.20 points on the PCL-5 compared to 7.77 points in the Wait-list group; Effect size (Cohen's d) = -0.75, 95% CI 2-sided [-1.85 to 0.35]

2. Secondary Outcome: Change in Total Score on the Clinician-Administered PTSD Scale for DSM-5 (CAPS)
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS) is a semi-structured interview that assesses the severity of current symptoms for Posttraumatic Stress Disorder (PTSD). The total score ranges from 0 (no symptoms) to 80 (maximal symptoms).
Time Frame: Baseline and 3-month follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months
Number analyzed (Participants) | 9 | 10
units on a scale | 1.4 (3.0) | 1.5 (2.9)
Statistical Analysis 1: Comparison: Shelter Dog Adoption vs Wait-list, Then Adoption After 3 Months; Test type: Superiority; p = 0.982, effect size (Cohen's d); effect size (Cohen's d) = -0.0

3. Secondary Outcome: Change in Alcohol Use Disorders Identification Test (AUDIT-C) Total Score
Description: Self-rating scale that assesses the frequency and extent of hazardous drinking. The range of the scale is from 0 (no hazardous drinking) to 12 (extremely hazardous drinking).
Time Frame: Baseline and 3-month follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months
Number analyzed (Participants) | 9 | 10
units on a scale | -0.5 (0.6) | 0.7 (0.6)
Statistical Analysis 1: Comparison: Shelter Dog Adoption vs Wait-list, Then Adoption After 3 Months; Test type: Superiority; p = 0.160, effect size (Cohen's d); effect size (Cohen's d) = -0.5

4. Secondary Outcome: Change in Beck Depression Inventory - II (BDI-II) Score
Description: The Beck Depression Inventory - II is a self rating scale that assesses the severity of depressive symptoms. The range of the scale is from 0 (no symptoms) to 63 (maximal symptoms).
Time Frame: Baseline and 3-month follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months
Number analyzed (Participants) | 9 | 10
units on a scale | -6.41 (1.72) | -0.19 (1.50)
Statistical Analysis 1: Comparison: Shelter Dog Adoption vs Wait-list, Then Adoption After 3 Months; Test type: Superiority; p = 0.015, effect size (Cohen's d); effect size (Cohen's d) = -1.36, 95% CI 2-sided [-2.49 to -0.23]

5. Secondary Outcome: Change in Community Integration Questionnaire (CIQ) Total Score
Description: Self-rating scale that assesses the extent of a subject's integration into her or his community. The range of the scale is from 0 (minimal integration) to 29 (maximal integration). A positive change indicates an improvement in integration.
Time Frame: Baseline and 3-month follow-up visit
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months
Number analyzed (Participants) | 9 | 10
units on a scale | 2.9 (1.1) | 2.1 (1.0)
Statistical Analysis 1: Comparison: Shelter Dog Adoption vs Wait-list, Then Adoption After 3 Months; Test type: Superiority; p = 0.59, Mixed Models Analysis; effect size (Cohen's d) = 0.2

6. Secondary Outcome: Change in Patient Health Questionnaire-9 (PHQ-9) Score
Description: The Patient Health Questionnaire-9 (PHQ-9) is a self-rating scale that assesses the severity of the symptoms of a major depressive episode. Scores range from 0 (no symptoms) to 27 (maximal symptoms).
Time Frame: Baseline and 3-month follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months
Number analyzed (Participants) | 9 | 10
units on a scale | -4.07 (1.20) | 0.71 (1.13)
Statistical Analysis 1: Comparison: Shelter Dog Adoption vs Wait-list, Then Adoption After 3 Months; Test type: Superiority; p = 0.010, effect size (Cohen's d); mixed effects regression models = -1.41, 95% CI 2-sided [-2.50 to -0.31]

7. Secondary Outcome: Percent of Subjects Reporting More Frequent Physical Activity Sessions on the Physical Activity Questionnaire (PAQ)
Description: The PAQ is a self-rating scale that assesses the frequency and intensity of various types of physical activity over the previous 3 months. The percent reporting increased frequency of physical activity sessions can range from 0 to 100.
Time Frame: Baseline and 3-month follow-up
Measure: Number; unit: percent of participants
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months
Number analyzed (Participants) | 9 | 10
percent of participants | 40 | 33
Statistical Analysis 1: Comparison: Shelter Dog Adoption vs Wait-list, Then Adoption After 3 Months; Test type: Superiority; p = 0.13, Fisher Exact

8. Secondary Outcome: Change in the Global Score on the Pittsburgh Sleep Quality Inventory With PTSD Addendum (PSQI-A)
Description: Self-rating scale that assesses the frequency and severity of various sleep-related problems, including problems that frequently occur in persons with PTSD. Scores range from 0 (excellent sleep quality) to 42 (very poor sleep quality).
Time Frame: Baseline and 3-month follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months
Number analyzed (Participants) | 9 | 10
units on a scale | -1.3 (1.4) | 1.3 (1.2)
Statistical Analysis 1: Comparison: Shelter Dog Adoption vs Wait-list, Then Adoption After 3 Months; Test type: Superiority; p = 0.188, effect size (Cohen's d); effect size (Cohen's d) = 0.9

9. Secondary Outcome: Number of Participants With Improvement in Quality of Life After Dog Adoption
Description: Interview that asks open-ended questions to assess the subject's symptoms, quality of life, and experiences related to having a dog
Time Frame: Baseline and 1-month, 3-month, 4-month, and 6-month follow-up visits, as well as 2-week, 2-month, and 4.5-month phone calls
Population: Participants who had a dog for 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months
Number analyzed (Participants) | 6 | 4
Participants | 5 | 4

10. Secondary Outcome: Change in Scores on the UCLA Loneliness Scale, Version 3
Description: The UCLA Loneliness Scale, Version 3 is a self-rating scale that measures the severity of symptoms of loneliness. The range of the scale if from 20 (no symptoms) to 80 (maximal symptoms).
Time Frame: Baseline and 3-month follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months
Number analyzed (Participants) | 9 | 10
units on a scale | -7.8 (3.5) | 3.4 (3.3)
Statistical Analysis 1: Comparison: Shelter Dog Adoption vs Wait-list, Then Adoption After 3 Months; Test type: Superiority; p = 0.031, mixed effects regression models; effect size (Cohen's d) = 1.2

11. Secondary Outcome: Changes in the Mental Component Score of the Veterans RAND 12-item Health Survey (VR-12)
Description: The VR-12 is a12-item self-rating scale that assess health-related quality of life. The results are expressed as two scores, a Mental Component Score and a Physical Component Score. The Mental Component Score measures mental aspects of quality of life and ranges from 0 (extremely poor mental health) to 100 (extremely good mental health), while the Physical Component Score measures physical aspects of quality of life and also ranges from 0 (extremely poor physical health) to 100 (extremely good physical health).
Time Frame: Baseline and 3-month Follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months
Number analyzed (Participants) | 9 | 10
units on a scale | 6.01 (4.34) | 2.30 (4.06)
Statistical Analysis 1: Comparison: Shelter Dog Adoption vs Wait-list, Then Adoption After 3 Months; Test type: Superiority; p = 0.541, effect size (Cohen's d); effect size (Cohen's d) = 0.30, 95% CI 2-sided [-0.80 to 1.40]

12. Secondary Outcome: Changes in Current Pain Ratings on the Numeric Rating Scale for Pain Intensity (NPS)
Description: The NPS asks patients to rate their pain intensity on a scale from 0 (no pain) to 10 (worst possible pain)
Time Frame: Baseline and 3-month follow-up
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Shelter Dog Adoption: Veterans will choose a dog from the San Antonio Humane Society with the help of a San Antonio Humane Society adoption counselor and study staff and take it home to live with them. The dog will be a pet and not a service dog.
  Following adoption, Veterans and their dogs will receive 8 weeks of free obedience training provided by a veterinarian,
- Wait-list, Then Adoption After 3 Months: After 3 months on a wait-list, Veterans will choose a dog from the San Antonio Humane Society with the help of a San Antonio Humane Society adoption counselor and study staff and take it home to live with them The dog will be a pet and not a service dog. Following adoption, Veterans and their dogs will receive 8 weeks of free obedience training by a veterinarian.
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months
Number analyzed (Participants) | 9 | 10
units on a scale | -0.1 (0.7) | -1.6 (0.7)
Statistical Analysis 1: Comparison: Shelter Dog Adoption vs Wait-list, Then Adoption After 3 Months; Please note that a minus number indicates an increase in pain ratings; Test type: Superiority; p = 0.139, effect size (Cohen's d); effect size (Cohen's d) = 0.6

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Shelter Dog Adoption | Wait-list, Then Adoption After 3 Months
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 5/9 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shelter Dog Adoption (N=9) | Wait-list, Then Adoption After 3 Months (N=10)
Emotional distress - reasons given under Additional Description (Psychiatric disorders) | 5 (5) | 4 (6) — wished dog had more room to run, worried dog was at home alone, unhappy was assigned to wait-list, dog chewed up things, dog dug up yard, dog too energetic, dog smelled bad, dog growled (2), dog had medical problems (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No